CLINICAL TRIAL: NCT06627101
Title: Prevalence of Traditional Medicine Use in Patients With Chronic Low Back Pain in Northern Brazil: a Cross-sectional
Brief Title: Traditional Medicine Use in Low Back Pain
Acronym: TMLBP
Status: Not yet recruiting | Type: Observational
Sponsor: Federal University of Amapa (Other)
Responsible Party: Principal Investigator, Natalia Camargo Rodrigues Iosimuta, Professor, Federal University of Amapa
Other Study IDs: 7.010.322
Record Dates: First submitted 2024-09-26; First posted 2024-10-04 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: Traditional Medicine; Beliefs; Lower back pain.
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic low back pain (CLBP) is classified as one of the leading causes of disability worldwide. Furthermore, the painful experience of CLBP can be influenced by some already established factors, such as beliefs, self-efficacy, and kinesiophobia. Beliefs are pre-established ideas that can influence physical functionality, pain experience, social functioning, and adherence to CLBP treatment Clique ou toque aqui para inserir o texto. Among them is Traditional Medicine, a practice carried out by some populations that continue to trust their own popular medicine to meet their health demands. According to the WHO, Traditional Medicine (MT) or Popular Medicine (MP) is a practice reproduced in different cultures and based on beliefs, the sum of experiences and knowledge, whose objective is to prevent, treat or cure illnesses, whether physical or mental. This habit includes the use of home remedies, which are based on the manipulation of plant, animal, and mineral extracts for therapeutic purposes. Furthermore, it is important to point out that, as it is a chronic condition, individuals living with CLBP are strongly influenced by psychological factors, such as kinesiophobia (avoidance of exercise), catastrophizing (intensifying fear of movement, as they feel that pain is a threat), and low self-efficacy in processing and modulating pain, increasing levels of pain and disability. Also, in addition to this, socioeconomic level is one of the determinants of the incidence and intensity of chronic pain. In short, although the practice of TM has been recognized for decades, it is not known whether there is a relationship between this belief and the levels of self-efficacy, kinesiophobia and catastrophizing of individuals with CLBP in Northern Brazil. Therefore, this study aims to identify the use of TM and its impacts on the functional activities and quality of life of individuals with CLBP in the northern region of Brazil. This is a cross-sectional observational study. Individuals participating in this research will be invited to respond online to the questionnaire prepared by the authors of this study. Continuous data will be analyzed descriptively using mean and standard deviation; categorical data will be described in frequency form, and the normality of the data will be analyzed to identify the possibility of using parametric or non-parametric statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* individuals over 18 years of age
* both genders
* diagnosed with chronic low back pain
* who have had pain for at least three months
* who are natives of the Northern region of Brazil

Exclusion Criteria:

* Individuals with low back pain of oncological origin
* recent traumas that may have caused the pain (such as falls, car accidents, and fractures)
* patients in the postoperative period
* bedridden patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include individuals over 18 years of age, of both genders, diagnosed with chronic low back pain, who have had pain for at least three months, and who are natives of the Northern region of Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Estimated)
Dates: Start 2024-10-26 (Estimated); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
prevalence of Traditional Medicine | 1 day
  a practice still relied upon by certain populations that continue to trust their own folk medicine to address their health needs

SECONDARY OUTCOMES:
functionality | 1 day
  the Oswestry Disability Index (ODI) questionnaire will be used. The instrument can be self-administered or administered through an interview, consisting of a series of 10 questions that address pain intensity and difficulties in daily life activities.
Self-Efficacy Assessment | 1 day
  The Chronic Pain Self-Efficacy Scale (AEDC) will be used, validated in Brazil. It is a specific scale for measuring the perception of self-efficacy and the ability to cope with the consequences of pain in patients with chronic pain. It consists of 22 items divided into three factors or domains: self-efficacy for pain control (PSE), self-efficacy for physical function (FSE), and self-efficacy for symptom control (CSE). Each belief is assessed on a Likert scale ranging from 10 to 100, reflecting the certainty regarding each item

IPD SHARING:
Plan to Share IPD: No